CLINICAL TRIAL: NCT00587444
Title: Optimal Heparin Dosing Regimens for Cardiopulmonary Bypass
Acronym: Heparin Dosing
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Dr. William Oliver, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 330-01; 3300100; CR4023159908
Record Dates: First submitted 2007-12-21; First posted 2008-01-07 (Estimated); Last update posted 2009-10-15 (Estimated); Status verified 2009-10

CONDITIONS: Postoperative Hemorrhage
Keywords: heparin management
MeSH Terms: conditions — Postoperative Hemorrhage | interventions — Heparin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Other): control standard dose heparin dose
  Interventions: Drug: Heparin
- 2 (Active Comparator): high dose heparin dose
  Interventions: Drug: HH or high heparin
- 3 (Active Comparator): hepcon guided therapy
  Interventions: Drug: heparin concentration HC

INTERVENTIONS:
Drug: Heparin — 300u/kg of heparin for CPB ACT performed. If ACT is < 480 seconds a bolus of 5000u heparin will be given. ACT will be repeated and bolus given until ACT is>480 seconds
  Arms: 1
Drug: HH or high heparin — initial dose of 450u/kg for CPB ACT performed additional bolus given if result is <600 seconds anytime during CPB
  Arms: 2
Drug: heparin concentration HC — will have anticoagulation during CPB assessed with heparin concentration monitoring and heparin dose response (HDR) to determine the optimal dosage of heparin. This group will evaluate the possible benefit of the HDR to determine heparin dosing and monitoring to achieve maximal suppression of thrombin compared to a fixed dose of heparin as the other two groups. Additional heparin doses will be given to maintain a specific heparin concentration according to the HDR. This is a recognized way of managing heparin dosing and anticoagulation for CPB.
  All three groups will have heparin neutralized by protamine. Adequacy of heparin neutralization will be based on a difference between the ACT and heparinase-treated ACT values of less than 10%
  Arms: 3

SUMMARY:
Study has been completed and is in the data analysis and manuscript writing phase of the project.

ELIGIBILITY:
Inclusion Criteria:

* Adult male and non-pregnant female patients scheduled for elective cardiac surgery requiring CPB will be eligible for enrollment.

Exclusion Criteria:

* Age less than 18 or greater than 90 years; emergency surgery
* Circulatory arrest
* Combined non-cardiac procedures such as carotid endarterectomy
* Congenital heart repair
* Off-CPB coronary artery bypass grafting (CABG)
* Clotting disorder
* Fibrinolytic agents (e.g. streptokinase), severe hepatic disease
* Aprotinin use
* Cooling < 28 degrees C during CPB
* Dialysis dependent renal failure; and
* Platelet receptor GP3a/2b antagonists medication received within 48 hours of surgery. Patients that are not receiving tranexamic acid (TA) intraoperatively will be excluded.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2001-06; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
measure blood loss | within 48 hours

SECONDARY OUTCOMES:
transfusion requirements | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: William Oliver, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States